CLINICAL TRIAL: NCT04448613
Title: Precise High Resolution MRI to Increase Accuracy and Gain Confidence to Diagnose Patients With Optic Disc Edema
Acronym: PAGODE
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: 2020-A00502-37
Record Dates: First submitted 2020-06-22; First posted 2020-06-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Optic Disk; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI — Patients with optic disc swelling diagnosed by a fundus and included in the study will have a brain MRI and visual pathways lasting 30 minutes.
  Two additional 10-minute sequences will be added to the standard protocol.

SUMMARY:
The presence of optic disc swelling at the fundus is a non-specific clinical sign that can occur in many ophthalmologic, neuro-ophthalmologic or encephalic pathologies. The diagnostic range is vast, including inflammatory pathologies of the optic nerve, infiltrative or compressive orbital pathologies, idiopathic or secondary intracranial hypertensions, not to mention the pseudo optic disc swelling found in drüsens.

MRI is increasingly being used as a first-line examination to obtain an etiologic diagnosis in a patient with optic disc swelling. It allows a rapid diagnosis to be made in cases of inflammatory pathology or compressive or infiltrative pathology. It can provide very suggestive elements in the case of intracranial hypertension. It appears to be potentially useful in diagnosing ischemic optic neuropathy or in directing towards an etiological diagnosis of Giant Cell Arteritis.

The development of new high-resolution MRI sequences has made it possible to obtain extremely fine resolutions of a few hundred microns in the plane. Apart from a few clinical cases and small series, there is no precise evaluation of the interest of these new sequences in the positive and etiological diagnosis of ophthalmological, neuro-ophthalmological and encephalic pathologies responsible for the presence of optic disc swelling.

The objective of our study is therefore to evaluate the diagnostic contribution and the gain in diagnostic confidence provided by these new sequences in the context of pathologies manifesting as optic disc swelling.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* presenting a papillary edema detected clinically at the back of the eye
* Express consent to participate in the study
* Affiliate or beneficiary of a Social Security scheme

Exclusion Criteria:

* MRI contraindication (electrical device, metallic foreign body, claustrophobia)
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the radiology service of the A. de Rothschild foundation and presenting a papillary edema detected clinically at the back of the eye sent by the emergency department for an MRI
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
FLAIR hypersignal size: larger diameters and area | baseline
  larger diameters and area of FLAIR hypersignal

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild (FOR), Paris, France